CLINICAL TRIAL: NCT06281288
Title: Effect of Cognitive-Behavioral Therapy Combined With Exercise Training in Adolescent Females With Elevated Depression Symptoms
Brief Title: Cognitive-Behavioral Therapy With Exercise Training in Adolescent Females With Elevated Depression Symptoms
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Doaa Tammam Atia (Other)
Responsible Party: Sponsor-Investigator, Doaa Tammam Atia, Department of Physical Therapy for Pediatrics, Faculty of Physical Therapy, Suez University, P.O.Box:43221, Suez, Egypt, Suez University
Organization: Suez University (Other)
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Prevention
Other Study IDs: P.T.REC/012/004754
Record Dates: First submitted 2024-02-20; First posted 2024-02-28 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Cognitive Behavioral Therapy; Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- cognitive therapy with regular exercise (Experimental): In the form of regular exercise where each participant perform exercise training approximately 60-min 3 times per week for 12 weeks, each session includes a combination of moderate intensity (~63% maximum heart rate; HRmax) aerobic (~25 min) and resistance (~25 min) activities, with additional time for warm-up (5 min; 10% HRmax) and cool down (5 min).
  Interventions: Behavioral: Cognitive-Behavioral Therapy; Other: Exercise Training
- cognitive therapy with irregular exercise (Experimental): in form of irregular exercise training approximately 60-min once a week for 12 weeks, each session include a combination of moderate intensity (~63% maximum heart rate; HRmax) aerobic (~25 min) and resistance (~25 min) activities, with additional time for warm-up (5 min; 10% HRmax) and cool down (5 min).
  Interventions: Behavioral: Cognitive-Behavioral Therapy; Other: Exercise Training
- cognitive therapy only (Experimental): Cognitive behavioral therapy) CBT (techniques is co facilitated by a psychiatrist where participants attend 12 sessions during the 12 weeks of treatment. The intervention is 60-min weekly in group sessions
  Interventions: Behavioral: Cognitive-Behavioral Therapy

INTERVENTIONS:
Behavioral: Cognitive-Behavioral Therapy — Cognitive behavioral therapy
Other: Exercise Training — Moderate intensity (~63% maximum heart rate; HRmax) aerobic (~25 min) and resistance (~25 min) activities
  Arms: cognitive therapy with irregular exercise; cognitive therapy with regular exercise

SUMMARY:
PURPOSE: To Study the Effect of Cognitive-behavioral therapy combined with exercise training in adolescent females with elevated depression symptoms

BACKGROUND: Teenagers are more likely than any other age group to experience psychological issues due to depression, Adolescents have gotten active attention from society for their mental health difficulties since they are a high-level reserve talent stratum in society. Adolescent depression rates have increased in recent years, and "silent killers" are preying on them. Teenagers are more likely than any other age group to experience psychological issues due to depression, Adolescents have gotten active attention from society for their mental health difficulties since they are a high-level reserve talent stratum in society. Adolescent depression rates have increased in recent years, and "silent killers"

RESEARCH QUESTION: Is there is an effect of exercise on depression in adolescent girls.

DETAILED DESCRIPTION:
The interventions start after assessment of depression to know the level of depression by using the Center for Epidemiological Studies Depression Scale for Children (CES-DC), and the exercise intervention consist of physical activity combined with Cognitive behavioral therapy. Group - A perform regular physical activity in addition to cognitive therapy, Group - B perform irregular physical activity in addition to cognitive therapy, Group - C cognitive therapy only

ELIGIBILITY:
Inclusion Criteria:

* 1. Depression adolescent girls 2. All patients should be in school

Exclusion Criteria:

1. obesity
2. malignant diseases
3. psychotic disorders or psychosis.
4. Permanent long-term psychiatric medication

Ages: 12 Years to 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2023-12-25 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Center for Epidemiological Studies Depression Scale for Children (CES-DC), | First at baseline and then after 12 weeks of the exercise program
  is a 20-item self-report depression inventory with possible scores ranging from 0 to 60. Each response to an item is scored as follows: 0 = "Not At All" 1 = "A Little" 2 = "Some" 3 = "A Lot" However, items 4, 8, 12, and 16 are phrased positively, and thus are scored in the opposite order: 3 = "Not At All" 2 = "A Little" 1 = "Some" 0 = "A Lot" Higher CES-DC scores indicate increasing levels of depression.

CONTACTS AND LOCATIONS:
Overall Officials: Sally MS Mahmoud, Dr., Principal Investigator — Misr University for Science and Technology, Giza, Egypt.
Locations (1):
- doaa Tammam Atia, Suez, Egypt

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication would be available after the end of the study
Supporting Information: Study Protocol, CSR
Time Frame: 10 months
Access Criteria: requesting the main author